CLINICAL TRIAL: NCT00707499
Title: A Single-Dose, Phase I, Dosimetry, Biodistribution, and Safety Trial of BMS 747158 in Healthy Subjects
Brief Title: A Phase I Study in Healthy Volunteers to Assess Safety of BMS747158
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BMS747158-101
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2011-10

CONDITIONS: Healthy
MeSH Terms: interventions — BMS 747158-02

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: BMS747158

INTERVENTIONS:
Drug: BMS747158 — Single dose administration.

SUMMARY:
The purpose of this clinical research study is to learn the safety and biodistribution of BMS747158 in normal, healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* age 18-40
* BMI 18-30 kg/m2
* No active or chronic illnesses
* If female: not pregnant, use of birth control or not of child-bearing potential

Exclusion Criteria:

* Significant active or chronic illness
* Any neurological disorder
* GI disease within 3 months
* Recent infection
* Major surgery within 4 weeks
* Donation of blood within 4 weeks
* Blood transfusion within 4 weeks
* Recent history drug/alcohol abuse
* Head trauma
* Significant screening ECG, EEG, lab tests, physical exam and vital signs abnormalities
* Prescription or OTC drugs within 2 weeks
* Exposure to any other investigational drug/device within 6

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Dosimetry analysis following whole body imaging after resting injection | Imaging takes place 0 - 310 minutes post injection

SECONDARY OUTCOMES:
Safety analysis following vital signs, ECGs, EEG, neuro and physical exams, telephone and visit follow up, and blood draws for chemistry and hematology post injection of BMS747158 at rest | Screening (14 days prior to dosing) through 14 days post dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Jamshid Maddahi, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States